CLINICAL TRIAL: NCT01746290
Title: The PulsePoint Smartphone Application: Recruiting Bystanders to Provide Basic Life Support for Victims of Out-of-Hospital Cardiac Arrest
Brief Title: The PulsePoint Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The intervention (PulsePoint application) could not be implemented in Toronto as planned
Sponsor: Queen's University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Dr. Steven Brooks, Clinician-Scientist, Queen's University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 228304
Record Dates: First submitted 2012-11-12; First posted 2012-12-10 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Cardiac Arrest, cardiopulmonary resuscitation, automated external defibrillators, smartphones
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PulsePoint notification (Experimental): Conventional Emergency Dispatch PLUS The PulsePoint notification. In the event of a potential cardiac arrest identified by 911call-takers, data will be automatically pushed to PulsePoint smartphone application users within very close proximity to the emergency. This will be done in parallel with normal emergency dispatch of paramedics and fire fighters to the scene of the emergency. The activation radius around the emergency is somewhat variable, depending on phone signal strength, climate conditions and whether the phone is inside or outside, but is approximately 200-500 meters.
  Interventions: Other: PulsePoint notification
- Usual Care (No Intervention): Patients randomized to the control arm will receive conventional emergency medical dispatching procedures but no PulsePoint notification will be sent to nearby PulsePoint users.

INTERVENTIONS:
Other: PulsePoint notification — When the smartphone receives the alert data, the phone alarms with auditory, tactile (vibration) and visual stimuli (Figure 1). After acknowledgement of the alert by the user, the application presents a map and text information to direct the user to the exact location of the emergency. Using local AED registry data, the application can also reveal exact AED locations in the vicinity of the emergency
  Arms: PulsePoint notification

SUMMARY:
"Sudden cardiac arrest" occurs when someone's heart stops beating unexpectedly. Each year, more than 45,000 Canadians have a cardiac arrest. A bystander can do three things to improve survival: Call 911,start chest compressions and apply a defibrillator. Together, these actions can increase survival by up to 800%. The problem is that bystanders to cardiac arrest only provide CPR in about 3 of every 10 cardiac arrest cases and AED use in about 3 of every 100 cardiac arrest cases. There are many people in the community who are trained and willing to provide help for cardiac arrest victims such as off-duty paramedics, fire fighters, nurses, etc. When a cardiac arrest occurs in the city, it is likely that one of these people is nearby, but unaware of the emergency. The PulsePoint smartphone application enables these people to be notified by the local emergency 911 service when there is a cardiac arrest near to them. It can be freely downloaded to several common types of smartphones. When there is a cardiac arrest emergency, all nearby PulsePoint users are sent an alert from the 911 service. When the phones receive the alert, they ring, vibrate and display a text message saying "CPR NEEDED". The user's current location and the exact location of the cardiac arrest are then displayed on a map. Nearby public access AEDs are also indicated on the map. The smartphone users can then go to provide chest compressions and use an AED while paramedics are on their way. A video at www.pulsepoint.org shows how this works. The objective of the investigators is to measure whether the PulsePoint smartphone application increases bystander CPR or AED use for victims of cardiac arrest outside the hospital. This project will happen in the City of Toronto. The investigators have a plan to get as many people as possible to download the application, focusing on health care professionals who know CPR. The investigators will set up a webpage that helps people download the software to their phone. The investigators will randomize 911 calls to have a PulsePoint alert sent or not. The investigators will use statistical analysis to measure whether sending an alert to a smartphone increases the chances of bystander resuscitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 911 calls assigned MPDS code 09-E-01 (Suspected atraumatic cardiac arrest not breathing), and 09-E-02 (Suspected cardiac arrest, not breathing normally),
2. Out-of-hospital cardiac arrest as defined within the ROC Epistry Database

Exclusion Criteria:

1. Trauma (including burns) associated with cardiac arrest
2. Cardiac arrests occurring in prisons, etc
3. Patients not treated by paramedics because of a DNR order or signs of obvious death as per Ontario provincial paramedic medical directives (e.g. decapitation, decomposition, rigour mortis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Bystander Resuscitation | Patients will be followed for this outcome during the interval from 911 call to emergency medical services arrival, an expected average of 5 minutes
  Bystander Resuscitation is defined as the occurrence of a bystander performing cardiopulmonary resuscitation or applying an automated external defibrillator to the chest of the subject prior to the arrival of professional rescuers

SECONDARY OUTCOMES:
Bystander CPR | Patients will be followed for this outcome during the interval from 911 call to emergency medical services arrival, an expected average of 5 minutes
  The performance of cardiopulmonary resuscitation by a bystander to cardiac arrest prior to arrival of professional rescuers
Bystander AED use | Patients will be followed for this outcome during the interval from 911 call to emergency medical services arrival, an expected average of 5 minutes
  The use of an automated external defibrillator by a bystander prior to the arrival of professional rescuers. Automated external defibrillator use is defined as the application of the electrical pads of the machine to the chest of the victim.
Bystander AED shock | Patients will be followed for this outcome during the interval from 911 call to emergency medical services arrival, an expected average of 5 minutes
  The occurrence of a bystander applying an automated external defibrillator and then applying a defibrillatory shock to the chest of the victim
Return of Spontaneous Circulation | Patients are followed until death or discharge from the hospital, an expected average 30 days
  Return of spontaneous circulation, defined as any palpable pulse or measureable blood pressure.
Survival to hospital discharge | Patients are followed until death or discharge from hospital, an expected average of 30 days
  Survival of a patient to the point of discharge from the acute care hospital. Discharge may be to a residence or long term care facility.
Survival to hospital discharge with good functional outcome | Patients are followed unitl death or discharge from hospital, an expected average of 30 days
  The occurrence of a patient surviving to hospital discharge with a Modified Rankin Score of 0, 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Brooks, MD MHSc, Principal Investigator — Queen's University
Locations (1):
- Toronto Emergency Medical Services, Toronto, Ontario, Canada